CLINICAL TRIAL: NCT01455129
Title: Early Intervention With Tiotropium （Spiriva） in Chinese Patients With Chronic Obstructive Pulmonary Disease (COPD): a Randomized, Double-blind, Placebo-controlled, Parallel, Multicentre Trial
Brief Title: Tiotropium In Early Chronic Obstructive Pulmonary Disease Patients in China
Acronym: Tie-COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Boehringer Ingelheim (Industry); Rundo International Pharmaceutical Research & Development Co.,Ltd. (Industry)
Responsible Party: Principal Investigator, Nanshan Zhong, Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 205.467
Record Dates: First submitted 2011-09-21; First posted 2011-10-19 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; COPD; COPD exacerbation; treatment; tiotropium; anticholinergic; acute exacerbation of COPD (AECOPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tiotropium group (Active Comparator): 18 mcg tiotropium, once daily, inhaled by HandiHaler
  Interventions: Drug: Tiotropium
- placebo group (Placebo Comparator): matching placebo, once daily, inhaled by HandiHaler
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Tiotropium — 18 mcg tiotropium capsule, once daily, inhaled by HandiHaler, for 24 months
  Other Names: Spiriva
  Arms: tiotropium group
Drug: placebo — placebo, once daily, inhaled by HandiHaler
  Arms: placebo group

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is one of the commonest respiratory diseases. During the early stage of COPD, patients only have mild respiratory symptoms or signs which may lead to under-diagnosis of the disease. Patients may show poor response to treatment at later stages of the disease, associated with higher mortality and incidence of re-hospitalization and disability causing burden for both the families and the society.

So far, there is no large-scale clinical trial on long-term intervention with tiotropium bromide (Spiriva) in patients with early stages of COPD (i.e. GOLD Stage I-II COPD or asymptomatic COPD). It would be of great significance for COPD prevention and treatment if the investigators could prove that tiotropium decreases the lung function decline and reverses disease progression in patients with early-stage COPD.

The investigators objective is to evaluate the efficacy of long-term intervention with tiotropium in early stage (FEV1 ≥50% predicted) COPD (difference of trough FEV1, number of exacerbations, time to first exacerbation, quality of life, etc) and relevant pharmacoeconomic endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40-85 yrs, both male and female, with or without smoking history, receiving treatment in community hospitals or outpatient department in general hospitals
* GOLD Stage I-II COPD: FEV1/FVC<70% and FEV1≥50% predicted, measured 20min after 400μg salbutamol inhalation
* With stable COPD: no COPD exacerbation during the latest 4 weeks prior to the recruitment
* With capability of communicating via oral conversation or written documents and signing informed consent
* With agreement to receive and are capable of participating in study related auxiliary examinations
* Capability of proper use of HandiHaler

Exclusion Criteria:

* Significant diseases other than COPD. A significant disease is defined as a disease or condition which, in the opinion of the investigator, may put the patient at risk because of participation in the study or may influence either the results of the study or the patients' ability to participate in the study
* Patients with clinically significant abnormal baseline haematology, blood biochemistry or urinary analysis, if the abnormality defines a significant disease as defined in exclusion criteria No. 1
* Patients with clinical diagnosis of lung cancer, bronchiectasis, pneumoconioses, or other single restricted ventilation
* Severe cardiovascular, neural, hepatic, renal and hematologic diseases or malignancies that may interfere with the operation of the study
* Patients with prostatic hyperplasia or bladder neck obstruction with significant symptoms, or narrow angle glaucoma
* Patients with known moderate to severe impaired renal function in the opinion of the investigator or creatinine clearance ≤50 ml/min
* Patients with history of asthma, allergic rhinitis, or who have a blood eosinophil count ≥600/mm^3
* Patients with active pulmonary tuberculosis
* Patients with life-threatening pulmonary embolism, α1-antitrypsin deficiency, or cystic fibrosis
* History of pneumonectomy
* COPD exacerbation in 4 weeks prior to the first visit (V0), or hospitalization and/or antibiotic application and/or oral or intravenous glucocorticosteroids application is required during screening stage.
* Treated with one of the trial drugs during the 30 days or 6 half-lives prior to the first visit (V0), with the selection of the longer period
* Long-term oxygen therapy, frequent use of glucocorticosteroids orally or intravenously at unstable doses(i.e. less than six weeks on stable doses) or at doses in excess of the equivalent of 10 mg of prednisone/day, or long-term use of antibiotics
* Pregnancy, lactation or potential of pregnancy
* Planned hospitalization or blood donation during the trial
* Known hypersensitivity or intolerance to trial drugs
* History of chronic alcohol or drug abuse, or any other conditions that may impact compliance
* Involvement in other clinical studies at the same time

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 841 (Actual)
Dates: Start 2011-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
difference of trough FEV1 at 24 months from baseline | at 24 months

SECONDARY OUTCOMES:
difference of peak FEV1 at 24 months from baseline | at 24 months
trough (pre-bronchodilator) FEV1 at 1, 6, 12 and 18 months | at 1, 6, 12 and 18 months
quality of life (CAT and CCQ) | at 1, 3, 6, 9, 12, 15, 18 and 24 months
symptom scores (mMRC dyspnoea scale) | at 1, 3, 6, 9, 12, 15, 18 and 24 months
time to first COPD exacerbation | 24 months
number of COPD exacerbation | 24 months
severity of COPD exacerbation | 24 months
Application of rescue medications | 24 months
drop-out rate | 24 months
adverse events | 24 months
peak (post-bronchodilator) FEV1 at 1, 6, 12 and 18 months | at 1, 6, 12 and 18 months
Yearly rate of decline in trough FEV1 from 1 month until completion of double-blind treatment | 24 months
Yearly rate of decline in peak FEV1 from 1 month until completion of double-blind treatment | 24 months
Yearly rate of decline in trough FVC from 1 month until completion of double-blind treatment | 24 months
Yearly rate of decline in peak FVC from 1 month until completion of double-blind treatment | 24 months
Yearly rate of decline in trough FEV1/FVC from 1 month until completion of double-blind treatment | 24 months
Yearly rate of decline in peak FEV1/FVC from 1 month until completion of double-blind treatment | 24 months
interval of COPD exacerbation | 24 months
duration of COPD exacerbation | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Nanshan Zhong, Professor, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University; Pixin Ran, Professor, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (25):
- China (25):
  - Beijing Chao-Yang Hospital, Beijing, Beijing Municipality
  - Xinqiao Hospital, Chongqing, Chongqing Municipality
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong
  - Liwan Hospital,Guangzhou Medical College, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong
  - Guangdong No.2 Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Guangzhou Panyu Center Hospital, Guangzhou, Guangdong
  - Huizhou First Hospital, Huizhou, Guangdong
  - Wengyuan County People's Hospital, Shaoguan, Guangdong
  - The First People's Hospital of Shaoguan, Shaoguan, Guangdong
  - Shaoguan Iron and Steel Group Company limited Hospital, Shaoguan, Guangdong
  - Shenzhen Sixth People's Hospital, Shenzhen, Guangdong
  - The second people's Hospital,Zhanjiang, Zhanjiang, Guangdong
  - Affiliated Hospital of Guangdong Medical College, Zhanjiang, Guangdong
  - The Affiliated Hospital of Guiyang Medical College, Guiyang, Guizhou
  - Guizhou People's Hospital, Guiyang, Guizhou
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Tongji Hospital,Tongji Medical College of HUST, Wuhan, Hubei
  - The Second People's Hospital of Hunan Province, Changsha, Hunan
  - Chenzhou No.1 people's Hopital, Chenzhou, Hunan
  - Shanghai Xuhui District Central Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Wu F, Dai C, Zhou Y, Deng Z, Wang Z, Li X, Chen S, Guan W, Zhong N, Ran P. Tiotropium reduces clinically important deterioration in patients with mild-to-moderate chronic obstructive pulmonary disease: A post hoc analysis of the Tie-COPD study. Respir Med. 2024 Feb;222:107527. doi: 10.1016/j.rmed.2024.107527. Epub 2024 Jan 8. PMID 38199288
- [Derived] Zhou Y, Zhong NS, Li X, Chen S, Zheng J, Zhao D, Yao W, Zhi R, Wei L, He B, Zhang X, Yang C, Li Y, Li F, Du J, Gui J, Hu B, Bai C, Huang P, Chen G, Xu Y, Wang C, Liang B, Li Y, Hu G, Tan H, Ye X, Ma X, Chen Y, Hu X, Tian J, Zhu X, Shi Z, Du X, Li M, Liu S, Yu R, Zhao J, Ma Q, Xie C, Li X, Chen T, Lin Y, Zeng L, Ye C, Ye W, Luo X, Zeng L, Yu S, Guan WJ, Ran P. Tiotropium in Early-Stage Chronic Obstructive Pulmonary Disease. N Engl J Med. 2017 Sep 7;377(10):923-935. doi: 10.1056/NEJMoa1700228. PMID 28877027
- [Derived] Li X, Zhou Y, Chen S, Zheng J, Zhong N, Ran P. Early intervention with tiotropium in Chinese patients with GOLD stages I-II chronic obstructive pulmonary disease (Tie-COPD): study protocol for a multicentre, double-blinded, randomised, controlled trial. BMJ Open. 2014 Feb 18;4(2):e003991. doi: 10.1136/bmjopen-2013-003991. PMID 24549160